CLINICAL TRIAL: NCT05657535
Title: Pain Relief Effect of Low-intensity Continuous Ultrasound Stimulator for Patients Suffering From Knee Arthritis; A Single-arm Pilot Clinical Trial
Brief Title: Pain Relief Effect of Low-intensity Continuous Ultrasound Stimulator for Knee Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyu Jae Lee (Other)
Responsible Party: Sponsor-Investigator, Kyu Jae Lee, Professor, Wonju Severance Christian Hospital
Organization: Wonju Severance Christian Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMB-2022-7; 2019-51-0458 (Other Grant/Funding Number: Mailtech Co.)
Record Dates: First submitted 2022-12-08; First posted 2022-12-20 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Before and after of treatment in single group
Masking Description: No need of blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Other): Single treatment group for evaluation pain relief before and after LICUS treatment
  Interventions: Device: Low-intensity continuous ultrasound stimulator

INTERVENTIONS:
Device: Low-intensity continuous ultrasound stimulator — Stimulation 5 minutes, 3 times a day for 4 weeks on the knee

SUMMARY:
The goal of this clinical trial is to test low-intensity continuous ultrasound stimulator(LICUS) for patients suffering from knee arthritis. it aims to evaluate the pain relief effect of LICUS.

35 participants were recruited, treated by LICUS on the knee joint for 5 minutes, 3 times a day for 4 weeks.

This study has single group and is for a before and after comparison of clinical treatment.

DETAILED DESCRIPTION:
Subject: 35 osteoarthritis patients Evaluation measure: Visual Analogue Scale (VAS), McMaster Universities Osteoarthritis Index (WOMAC) Method: A total of 35 subjects were selected in consideration of the dropout rate of 20%. Selected subjects were treated as a single group without randomization, and an appropriate amount of gel was applied to the knee OA pain area for 4 weeks. A blinded evaluation at baseline and after treat-ment was made. Primary outcome was pain on movement assessed by the VAS index. Secondary outcomes consisted of the WOMAC scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 to 60 years with pain due to OA of the knee and able to walk voluntarily
* Those who have more than one osteophyte in the tibiofemoral joint on radiographic findings (Kellgren-Lawrence gradesⅡ,Ⅲ)
* At visit 1 (screening) and visit 2, the pain status during knee OA activity was 100 mm pain VAS, as a result, those who are over 40mm
* If the Kellgren & Lawrence Grades are the same, target the one with the higher 100mm pain VAS
* Patients who are willing or able to follow the doctor's instructions, including joint movements
* Persons who can comply with concomitantly permitted drugs, prohibited drugs, and relief drugs
* Persons who can maintain the same exercise and activity during the clinical trial period
* Fully understand the purpose and procedure of this clinical trial

Exclusion Criteria:

* Those who have a history of rheumatoid arthritis or gouty arthritis or who have peripheral pain other than the knee joint patient.
* Those with fractures or dislocations on simple radiological examination.
* Those who are identified, or those with a similar risk of neuromuscular disease
* Those who have participated in other clinical trials within 6 months of participating in clinical trials.
* Patients with severe pain in the knee joint other than angular deformity, instability, and index knee in the knee joint
* Patients with other tumors other than degenerative knee arthrosis
* Persons with systemic symptoms that may affect knee pain
* Pregnant and lactating women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale(VAS) | 4 weeks
  Evaluation of pain on movement assessed by the VAS index

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 4 weeks
  Evaluation of pain on movement assessed by the WOMAC

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Jae Lee, Ph.D., Principal Investigator — Department of Convergence Medicine, Wonju College of Medicine, Yonsei University
Locations (1):
- Wonju College of Medicine, Wŏnju, Ganwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No